CLINICAL TRIAL: NCT00223301
Title: A One-Year Prospective, Randomized, Placebo-Controlled, Double-Blind, Phase II/III Safety Trial of Combination Therapy With IFN Beta-1a (Avonex) and Mycophenolate Mofetil (Cellcept) in Early Multiple Sclerosis
Brief Title: Safety Study of Combination Therapy With Intramuscular Avonex and Oral Cellcept in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Roche Pharma AG (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Elliot Frohman, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1103-716
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mycophenolate Mofetil (cellcept)

SUMMARY:
1. To determine the safety and tolerability of oral Cellcept when used in combination with weekly intramuscular Avonex in early MS.
2. To document changes in exacerbation frequency,
3. To document the incidence of mild, moderate, and severe exacerbations in the treated groups (categorical analysis),
4. To document changes in the level of sustained disability as measured by the expanded disability status score (EDSS) and ambulation index (AI),
5. To document changes in quality of life measures,
6. To assess fatigue with the validated fatigue assessment inventory,
7. Neuroimmunological studies:At baseline, 6 and 12 months after treatment

DETAILED DESCRIPTION:
Design: Uni-center, double-blind, randomized, placebo-controlled study of Avonex + placebo vs Avonex + Cellcept

Rationale: A number of immunopathogenic mechanisms have been hypothesized to figure prominently in the processes that culminate in the characteristic plaque lesion. These include the role of cytokines, chemokines, excitatory amino acids, free radicals, superoxides, and nitric oxide synthetase products. Recognizing that the disease process in MS involves a cascade of biological events, sets the stage for strategically targeting specific immunopathogenetic steps through rational combination therapy regimens. We now propose a combination clinical trial utilizing Avonex and mycophenolate mofetil (MMF), a novel agent with a broad spectrum of anti- inflammatory mechanisms.

* Study population: MS patients who have been diagnosed with clinically definite, laboratory supported definite, or monosymptomatic MS meeting CHAMPS criteria ref , of either sex, who are between the ages of 21 and 50 inclusive.
* Treatment Groups: 12 patients in each group, ALL patients on Intramuscular Avonex. Cellcept/Placebo will be started at 250mg bid for one week and then escalated by 250mg bid until a target dose of 1000mg bid is achieved and Avonex 30 mcg IM q week

Patients also see an examining physician every three months, have brain MRI scans done every other month and donate WBCs through a procedure called leukapheresis (done every six months).

* Efficacy Parameters/Evaluations: EDSS, PSAT, MSFC and MRI, relapse rate and safety measures
* Safety Parameters/Evaluations: Safety will be assessed by virtue of changes in T2/FLAIR lesions (number and volume) and in gadolinium enhancements (measured at 6 and 12 months after treatment initiation) compared to baseline measurements derived from one pretreatment run- in scan. In addition, a variety of clinical assessments will be performed for the period of 12 months of treatment. We will enroll 12 patients in each group (24 total)

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 21-45 inclusive
2. Clinically definite, laboratory supported definite relapsing MS of less than or equal to two years in duration or monosymptomatic MS meeting CHAMPS criteria ref .
3. At least one exacerbation in the preceding two years
4. Written informed consent.

Exclusion Criteria:

1. Primary progressive, secondary progressive or progressive relapsing MS.
2. Corticosteroids during the 60 days prior to study entry.
3. Treatment with plasma exchange within 90 days of preenrollment.
4. No prior exposure to total lymphoid irradiation.
5. No prior use of interferons, monoclonal antibodies, glatiramer acetate, methotrexate or other immunomodulatory drugs
6. A clinical relapse within 60 days prior to enrollment.
7. Pregnant/breastfeeding.
8. Patients with major medical illnesses.
9. Cognitive impairment interfering with ability to comply with the protocol.
10. Patients who need to remain on any contraindicated medication.
11. Diabetic
12. Inability to undergo MRI scan
13. On intravenous immunoglobulin protocol
14. HIV+ or RPR+
15. Females of childbearing age who have not undergone a sterilization procedure must be willing to practice effective birth control.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this safety/mechanistic study is to determine the safety and tolerability of oral Cellcept when used in combination with weekly intramuscular Avonex in early MS. Early MS for this study is defined at a definite diagnosis of less

SECONDARY OUTCOMES:
To document changes in exacerbation frequency
To document the incidence of mild, moderate, and severe exacerbations in the treated groups.
To document changes in the level of sustained disability as measured by the expanded disability status score (EDSS) and ambulation index (AI) as assessed by the Kaplan-Meier methodology.
To document changes in quality of life measures (MSQOL-54, SF-36, and Beck's Depression Index).
To assess fatigue with the validated fatigue assessment inventory
Neuroimmunological studies:At baseline, 6 and 12 months after treatment.
Pharmacodynamics.
Genetic Studies.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Frohman, MD/PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States